CLINICAL TRIAL: NCT05315154
Title: Sentinel Lymph Node Biopsy Versus No Axillary Surgery in Early Breast Cancer Clinically and Ultrasonographically Node-negative
Brief Title: Sentinel Lymph Node Biopsy Versus No Axillary Surgery in Early Breast Cancer
Acronym: VENUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Giuliano Mendes Duarte, MD PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06805118.2.1001.5404; RBR-8g6jbf (Registry Identifier: ReBEC)
Record Dates: First submitted 2022-03-20; First posted 2022-04-07 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No axillary surgery (Experimental)
  Interventions: Procedure: No axillary surgery
- Sentinel lymph node biopsy (Active Comparator)
  Interventions: Procedure: SLNB

INTERVENTIONS:
Procedure: No axillary surgery — In the study arm will be omitted surgery in axilla
  Arms: No axillary surgery
Procedure: SLNB — in the control arm will be realized SLNB
  Arms: Sentinel lymph node biopsy

SUMMARY:
The VENUS trial is a prospective, multicenter, noninferiority, randomized, controlled clinical trial that compares sentinel lymph node biopsy versus no axillary surgery in women with early breast cancer (tumor <5cm) and node-negative after clinical palpation and axillary ultrasound.

DETAILED DESCRIPTION:
The standard approach to women with early breast cancer (BC) and clinically negative nodes is sentinel lymph node dissection (SLND). Studies showed that axillary lymph node dissection (ALND) can be safely omitted in presence of positive sentinel lymph node in patients treated with breast conserving therapy.Therefore, the pertinence of SLND in the approach to women with early BC is being questioned, once it is not injury-free.

The ACOSOG Z0011 trial examined the safety of omitting ALND in patients with early BC and up to 2 positive nodes at SLND, undergoing conservative surgery plus breast radiotherapy. The 10-year worth of data from this trial strongly suggested that omitting the procedure in these restrict, well-selected, subsets of patients maybe safe. Neoadjuvant chemotherapy (NAC) may be the starting treatment step for women with aggressive BC subtypes even in early stages.The SENTINA and ACOSOG Z1071 trials revealed that for women with three or more negative nodes in SLND, the procedure's accuracy and false-negative rate lie within acceptable boundaries. Our hypothesis is that for patients with early BC (regardless of neoadjuvant systemic therapy), with clinically and ultrasound negative axilla, avoiding SLND may be safe from the oncological perspective.The VENUS trial will investigate whether there may be still room for further de-escalation of the approach to the axilla in well-selected subsets of BC patients, by including women for whom the de-escalation has not been tested in previous trials dealing with the subject.

The VENUS trial is a prospective, noninferiority, multicenter, randomized controlled clinical trial that was approved by the Local Research Ethic Committee .The trial will compare SLND with no axillary surgery in women with T1-2 invasive BC and N0 disease, as ascertained after clinical palpation and axillary ultrasound. Mastectomy and primary systemic therapy are allowed whether node negative previous start the treatment . All women accrued to the trial must sign the informed consent. Randomization 1:1 will be stratified by age (≤50 and >50 years old) and clinical tumor size (≤2 cm and >2 cm).

The sample size estimated is 364 women in each arm (400 to account for losses to follow-up). Sample size was calculated according to the following parameters: 90% disease-free survival in patients undergoing SLND and a minimum 85% in those not undergoing the procedure, 80% power and 95% confidence intervals, with a tolerated risk ratio of 0.8. After surgery, regardless of adjuvant therapies, and for at least 48 months, patients will undergo physical examination of their breasts and axilla every 6 months and mammography will be performed annually or at closer intervals if indicated. Adjuvant chemotherapy and radiotherapy will be performed according to the protocol of each participating center and patients without axillary surgery should be considered N0 for decision making.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 18 years or older
* Histologically confirmed invasive breast carcinoma (core or open biopsy), independent of hormone receptor and HER2 status
* Tumor smaller than 5 cm (T1 or T2) in clinical and radiological exams
* Clinically negative axilla
* Sonographically negative axilla or negative core biopsy/ fine needle biopsy (FNB) when ultrasound is suspect (lymph node tissue is required in core/FNB sample)
* Planned breast conservative surgery or mastectomy
* Written informed consent

Exclusion Criteria:

* Previous diagnostic of any invasive neoplasia (excluded skin cancer no melanoma)
* Metastatic disease in biopsy or image before treatment
* Withdrawal from participating of the study
* Initiated treatment for current breast cancer prior to study enrollment
* Pregnancy
* Breastfeed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-10-02 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 5 years
  Interval between the end of treatment and the diagnosis of any disease recurrence (breast, axilla or distant) by image exams or biopsy

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Defined time period between the end of treatment and the patient's death from any cause.
Locoregional free survival | 5 years
  Interval between the end of treatment and the diagnosis of any recorrence locoregional (breast or axilla) by biopsy
Axillary recurrence rate | 5 years
  Percentage of patients with disease recurrence in axilla by biopsy in each grup

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano Duarte, MD, PhD, Principal Investigator — Universidade Estadual de Campinas, Unicamp
Locations (18):
- Brazil (18):
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Maternidade Dona Iris, Goiânia, Goiás
  - Universidade Federal de Goiás, Goiânia, Goiás
  - Hospital de Clínica da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital do Câncer de Muriaé da Fundação Cristiano Varella, Muriaé, Minas Gerais
  - Universidade Federal do Paraná, Curitiba, Paraná
  - Hospital Barão de Lucena, Recife, Pernambuco
  - Oncocenter, Teresina, Piauí
  - Universidade Federal do Piauí, Teresina, Piauí
  - Hospital Federal da Lagoa, Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Hospital de Clínicas de Porto Alegre - UFRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor - Fundação Pio XII, Barretos, São Paulo
  - Unesp, Botucatu, São Paulo
  - Hospital Celso Pierro - PUCC, Campinas, São Paulo
  - Hospital da Mulher Prof.Dr. J A Pinotti - UNICAMP, Campinas, São Paulo
  - Hospital da Mulher, São Paulo, São Paulo
  - Hospital do Servidor Público Estadual, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo DCM, Duarte GM, Jales RM, Shinzato JY, Cardoso Filho C, Torresan RZ, Brenelli FP, Esteves SCB, Sarian LO. Sentinel lymph node biopsy vs no axillary surgery in early breast cancer clinically and ultrasonographically node negative: A prospective randomized controlled trial-VENUS trial. Breast J. 2020 Oct;26(10):2087-2089. doi: 10.1111/tbj.13994. Epub 2020 Jul 30. No abstract available. PMID 32729181
- [Background] Duarte GM, Araújo DCM, Jales RM, Shinzato JY, Cardoso Filho C, Torresan RZ, Brenelli FB, Kraft MBPL, Esteves SCB, Sarian LOZ, Rahal RMS, Freitas Jr R, Pessoa EC, Lucena CEM, Damin APS, Biazus JV, Budel VM, Oliveira Jr I, Vieira RAC, Gomes JCN. Sentinel lymph node biopsy versus no axillary surgery in early breast cancer clinically and ultrasonographically node negative: A multicentre prospective randomized controlled trial (VENUS trial. Cancer Research. 2022 82 (4_Supplement): OT1-04-03. DOI: https://doi.org/10.1158/1538-7445.SABCS21-OT1-04-03 Published: 15 February 2022